CLINICAL TRIAL: NCT03141372
Title: Urinary Retention Rates After Immediate Removal of Foley Catheter Versus Backfill Void Trial Following Total Laparoscopic Hysterectomy: A Randomized Controlled Trial
Brief Title: Urinary Retention After Total Laparoscopic Hysterectomy With Immediate Foley Catheter Removal Versus Backfill Void Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sara Farag (Other)
Responsible Party: Sponsor-Investigator, Sara Farag, Clinical Fellow in Minimally Invasive Gynecologic Surgery, Cleveland Clinic Florida
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FLA 17-020
Record Dates: First submitted 2017-05-03; First posted 2017-05-05 (Actual); Results first posted 2018-10-11 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Urinary Retention; Voiding Disorders
Keywords: Total Laparoscopic Hysterectomy; Urinary Retention; Backfill Void Trial; Autofill Void Trial
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to a backfill void trial following total laparoscopic hysterectomy or an autofill void trial following total laparoscopic hysterectomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Autofill Void Trial (Active Comparator): Patients who randomize to the autofill void trial will be allowed to urinate at any time within the first 3 hours after surgery. The amount urinated will be recorded using a commode specimen collection measurer. The PVR will be measured. If PVR > 100 mL, the void trial will be considered "failed" and a Foley catheter will be replaced.
  Interventions: Device: Void Trial using Foley catheter
- Backfill Void Trial (Active Comparator): About 300 mL of fluid will be instilled into the bladder and the Foley will then be removed. The participant will be given up to 1 hour to urinate and the amount urinated will be recorded using a commode specimen collection measurer. The PVR will be measured. If PVR > 100 mL or if the patient is unable to void within the hour, the void trial will be considered "failed" and a Foley catheter will be replaced.
  Interventions: Device: Void Trial using Foley catheter

INTERVENTIONS:
Device: Void Trial using Foley catheter — A void trial is a test to ensure that a subject does not have urinary retention after a surgical procedure. In an autofill void trial, the subject is allowed to void after surgery and the amount of resulting urine and the amount of urine still remaining in the bladder are measured. In a backfill void trial, water is instilled into the bladder, the foley is removed, and the subject is then allowed to urinate. Again, the amount of urine resulting and the amount of urine still in the bladder are measured.
  Other Names: Bladder challenge

SUMMARY:
Acute urinary retention is a complication of hysterectomies that can result in bladder over-distension and long term bladder dysfunction. The incidence of acute urinary retention after total laparoscopic hysterectomy (TLH) has been reported to be anywhere between 4% and 34%. Studies have varied in the method of post-operative bladder challenge and the modality of hysterectomy included. Moreover, most of the published studies are retrospective chart reviews or prospective observational studies, with a lack of randomized controlled trials. Risk factors for urinary retention include type of anesthesia used, how the hysterectomy is performed, use of post-operative narcotics, pre-operative urinary retention, and possibly aggressive bladder dissection. With the increased trend towards same-day discharge following TLH, urinary retention may cause unnecessary patient distress and a worsened post-operative course. Standardization of post-hysterectomy bladder challenge and identification of risk factors for urinary retention may aid in preventing urinary retention or acute bladder dysfunction. The primary objective is to compare the rate of void trial failure after TLH with the backfill technique versus the autofill technique.

DETAILED DESCRIPTION:
This will be a randomized control trial. Patients undergoing total laparoscopic hysterectomy (TLH) for benign conditions will be invited and consented to participate in the study prior to the day of their surgery. Each patient will be contacted by one of the study investigators and presented with the study including the risks, benefits, and follow up requirements. She will be given the option to participate and if agrees, she will sign a consent form. All enrolled participants will have a post-void residual (PVR) checked and recorded in the clinic using the bladder scanner that is available to us. The enrolled participants will also be asked to complete the Patient Perception of Bladder Condition (PPBC) and the Incontinence Impact Questionnaire-Short Form (IIQ-7) and the completed forms will be collected by the research team (see attached "Preoperative participant questionnaire").9,10 Each consented participant will be randomized to receive a post-operative backfill void trial or an autofill void trial on the day of her surgery. The participant will not be told of her randomization group pre-operatively; however, the surgical team will be aware of the randomization.

On the surgical day, all enrolled participants will undergo standard registration and preoperative preparation by the staff pre-operative nurse, including placement of intravenous access line and administration of standard preoperative medications. Preoperative medications (unless contraindicated due to allergy or other medication interaction) include single dose prophylactic antibiotics given prior to surgical incision, Tylenol 1,000 mg PO, Dexamethasone 10 mg IV (unless the participant has diabetes), Celebrex 200 mg PO (unless patient has a sulfa allergy, is ≥ 65 years old, weighs ≥ 50 kg, or has a CCl >50ml/min), Ondansetron 4 mg IV, and Gabapentin 600 mg PO (300 mg PO if participant is ≥ 65 years old) given in the preoperative area.11,12 Participants with a preoperative Caprini score of 5 or greater will also receive Heparin 5000 units subcutaneously for deep vein thrombosis (DVT) prophylaxis.13 The participant will be taken to the operating room. Induction, intubation, and anesthesia will be administered according to standard practice by a dedicated group of anesthesia providers. Prior to surgical incision, preoperative prophylactic antibiotics will be administered. The participant will be positioned in the dorsal lithotomy position with the lower extremities in the Allen stirrups bilaterally and the bilateral upper extremities in a tucked position. Surgical sterile preparation and draping will be performed per usual technique. Vaginal antiseptic preparation will be performed with 10% Povidone-Iodine solution. A Foley catheter will be placed prior to the start of the surgical procedure. The hysterectomy will then proceed in the usual manner. After the specimen is removed from the pelvis and the vaginal cuff is closed, a cystoscopy may be performed at the discretion of each surgeon. At this time, the randomization envelope will be opened. Participants who randomize to the backfill void trial will remain with a Foley catheter in place or will have the Foley catheter replaced, in the case that a cystoscopy is performed. Patients who randomize to the autofill void trial will be given a 500 cc bolus of crystalloid by the anesthesia team prior to leaving the operating room. All skin incisions will be closed in a subcuticular fashion and sealed with skin adhesive.

The participant will emerge from anesthesia under routine monitoring and will be transferred to the post-anesthesia care unit (PACU) when meeting appropriate criteria per anesthesia discretion. A staff PACU nurse will care for the participant in the PACU administer narcotic medications as necessary and/or per participant request. Once the participants are awake and meeting criteria for discharge, the patients in the backfill group will undergo a void trial by a PACU nurse or by a doctor if the nurse is unavailable. About 300 mL of fluid will be instilled into the bladder and the Foley will then be removed. The participant will be given up to 1 hour to urinate and the amount urinated will be recorded using a commode specimen collection measurer. The PVR will be measured using a bladder scanner. If the PVR is greater than 100 mL or if the patient is unable to void within the hour, the void trial will be considered "failed" and a Foley catheter will be replaced.

The participants in the autofill void trial group will be allowed to urinate at any time within the first 3 hours after surgery. The amount urinated will be recorded using a commode specimen collection measurer. The PVR will be measured using a bladder scanner. If the PVR is greater than 100 mL, the void trial will be considered "failed" and a Foley catheter will be replaced. We anticipate that most of these patients will void spontaneously within 2 hours of arrival to the PACU. At two hours post-operatively, any patient who cannot void or does not have the urge to void will have a bladder scan. If the patient has more than 300 cc in the bladder, she will be allowed 1 more hour to void. If she cannot, a Foley catheter will be placed and she will be considered to have failed the void trial. If the patient has less than 300 cc in the bladder, another 500 cc of crystalloid bolus will be given and we will await void for another hour. At 3 hours post-operatively, these patients will undergo another bladder scan. Those with greater than 300 cc of urine in the bladder will receive a Foley catheter. Those with less than 300 cc of urine in the bladder will have a backfill void trial by placing the remaining amount of fluid into the bladder for a total volume of 300 cc. The rest of the void trial will be completed as per normal backfill void trial protocol.

The participants who have a replaced Foley catheter will receive education regarding usage of a leg bag and will be discharged home to return to the office the following business day where a repeat void trial will be performed using the backfill method as previously outlined. If participants are unable to be discharged home, they will be admitted overnight in the hospital with documented rationale. A backfill void trial will then be performed the following day. If participants fail the 2nd void trial, a Foley catheter will be replaced and will remain in place for 1 week, at which time a backfill void trial will be repeated once again in the office. If this void trial is failed as well, participants will be educated about and asked to perform self-catheterization at home and will follow up with Urogynecology.

All participants will be discharged home with uniform medication prescriptions and instructions for usage. The medications will include Ondansetron 4mg PO every 8 hours as needed for nausea/vomiting (quantity 12), Colace 100mg PO twice daily (quantity 60), scheduled Ibuprofen 600mg PO every 6 hours (quantity 30), scheduled Acetaminophen 650mg PO every 6 hours (quantity 30), and Oxycodone 5mg PO every 4 hours as needed for breakthrough pain (quantity 30). These prescriptions are based on recent anesthesia practice guidelines.14,15

At the post-operative visit 10-14 days after the surgery, the participants will be evaluated and examined in the office. They will be asked to complete a questionnaire which includes the IIQ-7, the PPBC, and a void trial satisfaction question (see attached "post-operative participant questionnaire"). Participants will also be asked if they obtained a Foley catheter outside of the hospital at any urgent care centers, other doctors' offices, or emergency rooms. Additionally, participants will be asked if they have any urinary problems including dysuria, hematuria, frequency, hesitancy, urgency, or incomplete emptying. If any urinary complaints exist, participants will be asked to provide a urine sample for testing by urinalysis and urine culture. Participants will be treated per physician preference. After treatment, participation in the study will be considered completed.

ELIGIBILITY:
Inclusion Criteria:

* Females at least 18 years of age
* Understand and voluntarily sign an informed consent form
* English-speaking (able to read and understand English)
* Undergoing total laparoscopic hysterectomy for benign indication

Exclusion Criteria:

* Undergoing concomitant procedures in addition to hysterectomy which may cause urinary dysfunction
* Undergoing robotic-assisted laparoscopy or laparotomy
* Known history of pre-operative urinary incontinence or retention
* History of prior bladder or prolapse surgery
* Neurologic or spinal cord injury affecting bladder function
* Pregnant women
* Evidence of gynecologic malignancy
* Currently taking anticholinergic medications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Sprague, MD, Principal Investigator — Cleveland Clinic Florida
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Won HR, Maley P, Chetty N, Chan K, Abbott J. Bladder dysfunction after gynecologic laparoscopic surgery for benign disease. J Minim Invasive Gynecol. 2012 Jan-Feb;19(1):76-80. doi: 10.1016/j.jmig.2011.09.013. Epub 2011 Nov 25. PMID 22118884
- [Background] Alessandri F, Mistrangelo E, Lijoi D, Ferrero S, Ragni N. A prospective, randomized trial comparing immediate versus delayed catheter removal following hysterectomy. Acta Obstet Gynecol Scand. 2006;85(6):716-20. doi: 10.1080/00016340600606976. PMID 16752265
- [Background] Ghezzi F, Cromi A, Uccella S, Colombo G, Salvatore S, Tomera S, Bolis P. Immediate Foley removal after laparoscopic and vaginal hysterectomy: determinants of postoperative urinary retention. J Minim Invasive Gynecol. 2007 Nov-Dec;14(6):706-11. doi: 10.1016/j.jmig.2007.06.013. PMID 17980330
- [Background] Liang CC, Lee CL, Chang TC, Chang YL, Wang CJ, Soong YK. Postoperative urinary outcomes in catheterized and non-catheterized patients undergoing laparoscopic-assisted vaginal hysterectomy--a randomized controlled trial. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Mar;20(3):295-300. doi: 10.1007/s00192-008-0769-6. Epub 2008 Nov 14. PMID 19009225
- [Background] Smorgick N, DeLancey J, Patzkowsky K, Advincula A, Song A, As-Sanie S. Risk factors for postoperative urinary retention after laparoscopic and robotic hysterectomy for benign indications. Obstet Gynecol. 2012 Sep;120(3):581-6. doi: 10.1097/AOG.0b013e3182638c3a. PMID 22914467
- [Background] Kandadai P, Saini J, Patterson D, O'Dell K, Flynn M. Urinary Retention After Hysterectomy and Postoperative Analgesic Use. Female Pelvic Med Reconstr Surg. 2015 Sep-Oct;21(5):257-62. doi: 10.1097/SPV.0000000000000151. PMID 25521470
- [Background] Foster RT Sr, Borawski KM, South MM, Weidner AC, Webster GD, Amundsen CL. A randomized, controlled trial evaluating 2 techniques of postoperative bladder testing after transvaginal surgery. Am J Obstet Gynecol. 2007 Dec;197(6):627.e1-4. doi: 10.1016/j.ajog.2007.08.017. PMID 18060956
- [Background] Geller EJ, Hankins KJ, Parnell BA, Robinson BL, Dunivan GC. Diagnostic accuracy of retrograde and spontaneous voiding trials for postoperative voiding dysfunction: a randomized controlled trial. Obstet Gynecol. 2011 Sep;118(3):637-642. doi: 10.1097/AOG.0b013e318229e8dd. PMID 21860294
- [Background] Uebersax JS, Wyman JF, Shumaker SA, McClish DK, Fantl JA. Short forms to assess life quality and symptom distress for urinary incontinence in women: the Incontinence Impact Questionnaire and the Urogenital Distress Inventory. Continence Program for Women Research Group. Neurourol Urodyn. 1995;14(2):131-9. doi: 10.1002/nau.1930140206. PMID 7780440
- [Background] Coyne KS, Matza LS, Kopp Z, Abrams P. The validation of the patient perception of bladder condition (PPBC): a single-item global measure for patients with overactive bladder. Eur Urol. 2006 Jun;49(6):1079-86. doi: 10.1016/j.eururo.2006.01.007. Epub 2006 Jan 24. PMID 16460875
- [Background] Nelson G, Altman AD, Nick A, Meyer LA, Ramirez PT, Achtari C, Antrobus J, Huang J, Scott M, Wijk L, Acheson N, Ljungqvist O, Dowdy SC. Guidelines for pre- and intra-operative care in gynecologic/oncology surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations--Part I. Gynecol Oncol. 2016 Feb;140(2):313-22. doi: 10.1016/j.ygyno.2015.11.015. Epub 2015 Nov 18. No abstract available. PMID 26603969
- [Background] Modesitt SC, Sarosiek BM, Trowbridge ER, Redick DL, Shah PM, Thiele RH, Tiouririne M, Hedrick TL. Enhanced Recovery Implementation in Major Gynecologic Surgeries: Effect of Care Standardization. Obstet Gynecol. 2016 Sep;128(3):457-66. doi: 10.1097/AOG.0000000000001555. PMID 27500337
- [Background] Caprini JA. Individual risk assessment is the best strategy for thromboembolic prophylaxis. Dis Mon. 2010 Oct;56(10):552-9. doi: 10.1016/j.disamonth.2010.06.007. No abstract available. PMID 20971324
- [Background] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847
- [Background] Urbach DR, Harnish JL, McIlroy JH, Streiner DL. A measure of quality of life after abdominal surgery. Qual Life Res. 2006 Aug;15(6):1053-61. doi: 10.1007/s11136-006-0047-3. PMID 16900285
- [Background] Boccola MA, Sharma A, Taylor C, Wong LM, Travis D, Chan S. The infusion method trial of void vs standard catheter removal in the outpatient setting: a prospective randomized trial. BJU Int. 2011 Apr;107 Suppl 3:43-6. doi: 10.1111/j.1464-410X.2011.10044.x. PMID 21492377
- [Background] Du J, Marshall D, Leyland J, Shaw L, Broome KE, Mason DF. Prospective, multicentre, randomized controlled trial of bladder filling prior to trial of void on the timing of discharge. ANZ J Surg. 2013 Apr;83(4):239-42. doi: 10.1111/j.1445-2197.2012.06253.x. Epub 2012 Sep 18. PMID 22984818
- [Background] Odom BD, Ehlert M, Gupta P, Cholyway R, Boura JA, Killinger KA, Sirls LT. Clinical Comparison of 2 Trial-of-Void Methods After Outpatient Midurethral Sling Placement. Female Pelvic Med Reconstr Surg. 2016 May-Jun;22(3):172-4. doi: 10.1097/SPV.0000000000000258. PMID 26945265
- [Background] Pulvino JQ, Duecy EE, Buchsbaum GM, Flynn MK. Comparison of 2 techniques to predict voiding efficiency after inpatient urogynecologic surgery. J Urol. 2010 Oct;184(4):1408-12. doi: 10.1016/j.juro.2010.05.096. Epub 2010 Aug 19. PMID 20727543
- [Background] Tunitsky-Bitton E, Murphy A, Barber MD, Goldman HB, Vasavada S, Jelovsek JE. Assessment of voiding after sling: a randomized trial of 2 methods of postoperative catheter management after midurethral sling surgery for stress urinary incontinence in women. Am J Obstet Gynecol. 2015 May;212(5):597.e1-9. doi: 10.1016/j.ajog.2014.11.033. Epub 2014 Nov 27. PMID 25434837
- [Background] Turner LC, Kantartzis K, Shepherd JP. Predictors of postoperative acute urinary retention in women undergoing minimally invasive sacral colpopexy. Female Pelvic Med Reconstr Surg. 2015 Jan-Feb;21(1):39-42. doi: 10.1097/SPV.0000000000000110. PMID 25185611
- [Derived] Farag S, Padilla PF, Smith KA, Zimberg SE, Sprague ML. Postoperative Urinary Retention Rates after Autofill versus Backfill Void Trial following Total Laparoscopic Hysterectomy: A Randomized Controlled Trial. J Minim Invasive Gynecol. 2021 Apr;28(4):829-837. doi: 10.1016/j.jmig.2020.07.013. Epub 2020 Jul 24. PMID 32712322

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Autofill Void Trial | Backfill Void Trial
Started | 42 | 42
Completed | 42 | 40
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Autofill Void Trial | Backfill Void Trial | Total
Number analyzed (Participants) | 42 | 40 | 82
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 46 [41.3 to 50] | 46 [42.8 to 50] | 46 [42 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 40 | 82
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 16 | 35
  White | 23 | 23 | 46
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 32.4 [25.5 to 35.9] | 28.8 [25.8 to 33.9] | 30.2 [25.8 to 35.2]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Void Trial Failure Rate
Description: The primary endpoint of this study will be to determine if the rate of void trial failure after total laparoscopic hysterectomy is different after the autofill method versus the backfill method.
Time Frame: post-operative day, about 4 hours post-surgery
Measure: Count of Participants; unit: Participants
Groups:
- Autofill Void Trial: Patients who randomize to the autofill void trial will be allowed to urinate at any time within the first 3 hours after surgery. The amount urinated will be recorded using a commode specimen collection measurer. The postvoid residual will be measured. If postvoid residual greater than 100 mL, the void trial will be considered "failed" and a Foley catheter will be replaced.
  Void Trial using Foley catheter: A void trial is a test to ensure that a subject does not have urinary retention after a surgical procedure. In an autofill void trial, the subject is allowed to void after surgery and the amount of resulting urine and the amount of urine still remaining in the bladder are measured. In a backfill void trial, water is instilled into the bladder, the foley is removed, and the subject is then allowed to urinate. Again, the amount of urine resulting and the amount of urine still in the bladder are measured.
- Backfill Void Trial: About 300 mL of fluid will be instilled into the bladder and the Foley will then be removed. The participant will be given up to 1 hour to urinate and the amount urinated will be recorded using a commode specimen collection measurer. The postvoid residual will be measured. If postvoid residual greater than 100 mL or if the patient is unable to void within the hour, the void trial will be considered "failed" and a Foley catheter will be replaced.
  Void Trial using Foley catheter: A void trial is a test to ensure that a subject does not have urinary retention after a surgical procedure. In an autofill void trial, the subject is allowed to void after surgery and the amount of resulting urine and the amount of urine still remaining in the bladder are measured. In a backfill void trial, water is instilled into the bladder, the foley is removed, and the subject is then allowed to urinate. Again, the amount of urine resulting and the amount of urine still in the bladder are measured.
Arm/Group | Autofill Void Trial | Backfill Void Trial
Number analyzed (Participants) | 42 | 40
Participants | 7 | 11

2. Secondary Outcome: Time to Discharge
Description: The time to discharge will be measured for each participant. This will be determined by calculating the time between arrival to the post-anesthesia care unit and the time of discharge using documentation from Epic and from the case report forms.
Time Frame: post-operative day, about 4 hours post-surgery
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Autofill Void Trial | Backfill Void Trial
Number analyzed (Participants) | 42 | 40
minutes | 176 [160.5 to 255.5] | 218 [180 to 265]

3. Secondary Outcome: Number of Patients With Urinary Retention
Description: After discharge, participants will be monitored for any encounters for urinary retention (in our hospital system) and will be asked at their 10-14 day post-operative visit if they had a Foley catheter placed outside the hospital. Additionally, any participant who fails their 2nd void trial will be noted. The incidence of urinary retention post-discharge will be determined using this data.
Time Frame: 10-14 days post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Autofill Void Trial | Backfill Void Trial
Number analyzed (Participants) | 42 | 40
Participants | 1 | 1

4. Secondary Outcome: Number of Participants With Post-Operative Urinary Tract Infection
Description: Any participant diagnosed with a culture-proven urinary tract infection will be noted.
Time Frame: up to 14 days post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Autofill Void Trial | Backfill Void Trial
Number analyzed (Participants) | 42 | 40
Participants | 2 | 1

5. Secondary Outcome: Quality of Bladder Function Using the Incontinence Impact Questionnaire
Description: The Incontinence Impact Questionnaire-7 will be used to determine if there are any changes to the participants' short term quality of life before and after surgery. The questionnaire includes 7 questions asking how the participant's bladder function has affected her:
  1. Ability to do household chores.
  2. Physical recreation
  3. Entertainment activities
  4. Ability to travel by car or bus more than 30 minutes from home
  5. Participation in social activities outside the home
  6. Emotional health
  7. Feeling frustrated
  The patient scores each of the questions using the following scale:
  0 - Not at all
  1. - Slightly
  2. - Moderately
  3. - Greatly
  The scores were added and divided by 7 to obtain an average score for each participant. Hence the range of scores is 0 to 3 with 0 being the best and 3 being the worst.
Time Frame: pre-surgery and 14 days post-surgery
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Autofill Void Trial | Backfill Void Trial
Number analyzed (Participants) | 42 | 40
scores on a scale | 0 [0 to 1.75] | 0 [0 to 0]

6. Secondary Outcome: Patient Perception of Bladder Condition Score
Description: The Patient Perception of Bladder Condition will be used to determine if there are any changes to the participants' perception of bladder function before and after surgery.
  In this questionnaire, the participant answers one question as follows:
  My bladder condition:
  0 - Does not cause me any problems at all
  1. - Causes me very minor problems
  2. - Causes me some minor problems
  3. - Causes me (some) moderate problems
  4. - Causes me severe problems
  5. - Causes me many severe problems
  The score was recorded for each patient. The range of possible scores were 0 to 5 with 0 being the best and 5 being the worst scores.
Time Frame: presurgery and at 10-14 days post-surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Autofill Void Trial | Backfill Void Trial
Number analyzed (Participants) | 42 | 40
score on a scale | 0 [0 to 1] | 0 [0 to 1]

7. Secondary Outcome: Number of Participants Satisfied or Very Satisfied With Void Trial Using 5 Point Lickert Scale
Description: Participant satisfaction level with the method of void trial will be collected at the 10-14 day post-operative visit and compared between the two methods of void trial.
Time Frame: at 10-14 days post-surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Autofill Void Trial | Backfill Void Trial
Number analyzed (Participants) | 42 | 40
Participants | 39 | 30

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Autofill Void Trial | Backfill Void Trial
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/40
Other Adverse Events (participants affected / at risk) | 0/42 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT03141372/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT03141372/Prot_SAP_001.pdf